CLINICAL TRIAL: NCT07116213
Title: Clinical Research on Moderately Hypofractionated Adaptive Postoperative Radiotherapy for High-Risk Endometrial Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaorong Hou (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Hou, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHART-EC
Record Dates: First submitted 2025-06-09; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer; Hypofractionated Dose; Radiotherapy, Adjuvant; Side Effects; Survival , Tumor
Keywords: endometrial cancer; Hypofractionated dose; Radiotherapy
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Moderately Hypofractionated Adaptive Radiotherapy (Experimental)
  Interventions: Radiation: Moderately Hypofractionated Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Moderately Hypofractionated Adaptive Radiotherapy — Moderately Hypofractionated Adaptive Postoperative Radiotherapy

SUMMARY:
1. Study Type: Single-center, single-arm, prospective study.
2. Sample Size: 20 patients with high-risk endometrial cancer were enrolled.
3. Treatment Procedure:

   The existing clinical oART (Online Adaptive Radiotherapy) workflow protocol for malignant tumors used in our department was applied.

   Procedures included simulation, target volume delineation, radiotherapy planning, and treatment delivery.

   External beam radiation therapy (EBRT) was delivered using moderate hypofractionation.

   If indicated, brachytherapy was performed after the completion of EBRT. When combined with chemotherapy, radiotherapy could be administered during chemotherapy intervals or after completion of chemotherapy.
4. Study Endpoints:

Primary Endpoint: Incidence of acute toxicity. Secondary Endpoints: 3-year failure-free survival (FFS) rate, incidence of chronic toxicity, quality of life (QoL), treatment costs, etc.

DETAILED DESCRIPTION:
Research Process

1. Baseline Assessment Includes medical history inquiry, physical examination, and relevant laboratory/imaging tests. Complete the pre-radiotherapy Quality of Life Scale.
2. Treatment Plan

External Beam Radiotherapy (EBRT): Utilize online adaptive radiotherapy technology to irradiate the vagina and pelvic lymph node drainage areas. Employ moderate fractionation. Prescription Dose: 40.05 Gy / 15 fractions, administered once daily, five times per week.

Brachytherapy: Commence after completion of EBRT. Utilize 3D intracavitary brachytherapy technology. Fraction Dose: 4-6 Gy, for a total of 2-3 fractions, administered with an interval of 1-2 days between fractions.

3. Follow-up Visits

1. During Radiotherapy: Monitor CBC weekly and Biochemistry Panel every 2 weeks. Perform radiotherapy-related toxicity assessment.
2. Post-Radiotherapy:

Timepoints: End of radiotherapy; 3 months post-radiotherapy; 6 months post-radiotherapy; then every 6 months thereafter, until 3 years post-radiotherapy.

Follow-up Content: Includes medical history inquiry, physical examination, and Quality of Life assessment; Laboratory/Imaging Tests.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18-70 years old.
* Performance Status :

ECOG score 0-2.

* Expected to comply with oART (Online Adaptive Radiotherapy) workflow.
* Initial Surgical Treatment :

Total hysterectomy and bilateral salpingo-oophorectomy ± Pelvic and/or para-aortic lymph node dissection/sampling or sentinel lymph node biopsy.

* Pathological Staging & Histology (per FIGO 2009):

Stage I :

Grade 3 endometrioid adenocarcinoma with superficial myometrial invasion and extensive LVSI (Lymphovascular Space Invasion).

Grade 2 endometrioid adenocarcinoma with deep myometrial invasion and extensive LVSI.

Grade 3 endometrioid adenocarcinoma with deep myometrial invasion. Stage II-IIIC1 : Endometrioid carcinoma. Stage I-IIIC1 : Serous carcinoma or clear cell carcinoma.

* Informed Consent :
* Patients and families fully understand the study protocol.
* Voluntarily participate and sign informed consent forms before enrollment

Exclusion Criteria:

* Prior Radiotherapy : History of abdominal or pelvic irradiation.
* Treatment Interval :

Without adjuvant chemotherapy: >12 weeks between surgery and radiotherapy initiation.

With adjuvant chemotherapy: >6 months between surgery and radiotherapy initiation.

* Malignancy History : Prior diagnosis of other malignancies.
* Pregnancy/Lactation : Pregnant or breastfeeding women.
* Active Infection : Fever or uncontrolled active infection.
* Inflammatory Bowel Disease (IBD) : History of IBD (regardless of activity status).
* Comorbidities : Severe conditions affecting trial compliance, including: Unstable cardiac disease requiring treatment, renal impairment, chronic hepatitis, poorly controlled diabetes, psychiatric disorders

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | <90 days after treatment initiation
  Toxicities occurring <90 days from radiotherapy initiation. Evaluated using CTCAE v5.0.

SECONDARY OUTCOMES:
3-year failure-free survival | From date of surgery to the 3 years after treatment initiation
  The time from treatment initiation until the occurrence of any treatment failure events.
Chronic Toxicity | ≥90 days after treatment initiation
  Toxicities occurring ≥90 days from radiotherapy initiation. Evaluated using the RTOG Late Morbidity Scoring Schema.
Quality of Life (EORTC QLQ-C30/EORTC QLQ-EN24) | From date of surgery to the 3 years after treatment initiation
  EORTC QLQ-C30: This is a core quality of life questionnaire developed by the EORTC, applicable to all cancer patients. Scores are standardized to a 0-100 scale. For functional scales and the global quality of life scale, higher scores indicate better functioning or quality of life. For symptom scales/single items, higher scores indicate more severe symptoms or problems.
  EORTC QLQ-EN24: This is a module specifically designed to assess symptoms and quality of life unique to endometrial cancer patients. It serves as a supplementary module to the QLQ-C30 and cannot be analyzed independently. Scores are standardized to a 0-100 scale. For symptom items, higher scores indicate a greater symptom burden. For function/satisfaction items, higher scores indicate better function or satisfaction.
Treatment Costs | Through radiotherapy completion, an average of 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leung E, Gladwish AP, Davidson M, Taggar A, Velker V, Barnes E, Mendez L, Donovan E, Gien LT, Covens A, Vicus D, Kupets R, MacKay H, Han K, Cheung P, Zhang L, Loblaw A, D'Souza DP. Quality-of-Life Outcomes and Toxic Effects Among Patients With Cancers of the Uterus Treated With Stereotactic Pelvic Adjuvant Radiation Therapy: The SPARTACUS Phase 1/2 Nonrandomized Controlled Trial. JAMA Oncol. 2022 Jun 1;8(6):1-9. doi: 10.1001/jamaoncol.2022.0362. PMID 35420695
- [Background] Maddah Safaei A, Esmati E, Gomar M, Akhavan S, Sheikh Hasani S, Malekzadeh Moghani M, Zamani N, Moshtaghi M, Malek M, Jafari F, Sharifian A, Kolahdouzan K. Hypofractionated versus standard chemoradiotherapy in the definitive treatment of uterine cervix cancer: interim results of a randomized controlled clinical trial. J Cancer Res Clin Oncol. 2024 Jan 20;150(1):20. doi: 10.1007/s00432-023-05563-8. PMID 38244105
- [Background] Cho WK, Park W, Kim SW, Lee KK, Ahn KJ, Choi JH. Postoperative Hypofractionated Intensity-Modulated Radiotherapy With Concurrent Chemotherapy in Cervical Cancer: The POHIM-CCRT Nonrandomized Controlled Trial. JAMA Oncol. 2024 Jun 1;10(6):737-743. doi: 10.1001/jamaoncol.2024.0565. PMID 38662364